CLINICAL TRIAL: NCT00839163
Title: ODIXa-DVTA Prospective, Randomized, Multinational, Multicenter, Partially Blinded, Parallel-group, Open-label Active Comparator Controlled Phase II Dose Finding and Proof of Principle Trial.
Brief Title: Oral Direct Factor Xa Inhibitor BAY59-7939 in Patients With Acute Symptomatic Proximal Deep Vein Thrombosis(ODIXa-DVT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11223; 2004-001083-43 (EudraCT Number); ODIXa-DVT (Other: Company Internal)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2014-10

CONDITIONS: Venous Thrombosis; Deep Vein Thrombosis
Keywords: Embolism and Thrombosis; Pulmonary embolism; Embolism; Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Embolism and Thrombosis; Pulmonary Embolism; Embolism; Thrombosis | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 4 (Experimental)
  Interventions: Drug: Xarelto (Rivaroxaban, BAY59-7939)
- Arm 5 (Active Comparator)
  Interventions: Drug: Enoxaparin/Vitamin K-Antagonist

INTERVENTIONS:
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 10 mg bid main treatment period of 21 days followed by an extended period of trial therapy until week 12 (Day 84).
  Arms: Arm 1
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 20 mg bid main treatment period of 21 days followed by an extended period of trial therapy until week 12 (Day 84).
  Arms: Arm 2
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 30 mg bid main treatment period of 21 days followed by an extended period of trial therapy until week 12 (Day 84).
  Arms: Arm 3
Drug: Xarelto (Rivaroxaban, BAY59-7939) — 40 mg od main treatment period of 21 days followed by an extended period of trial therapy until week 12 (Day 84).
  Arms: Arm 4
Drug: Enoxaparin/Vitamin K-Antagonist — Enoxaparin/Vitamin K-Antagonist main treatment period of 21 days followed by an extended period of trial therapy until week 12 (Day 84). Enoxaparin was to be administered 1mg/kg bid sc for about 5-7 days. It was to be discontinued when INR was within the therapeutic range 2-3 for 2 consecutive days
  Arms: Arm 5

SUMMARY:
The purpose of this study is to compare the safety and efficacy of BAY59-7939 with the safety and efficacy of the licensed drug enoxaparin and a licensed oral vitamin K-antagonist and to find the optimal dose of BAY59-7939 for the anticipated phase III trials and for the future clinical use.

ELIGIBILITY:
Inclusion Criteria:

- Patients with acute symptomatic proximal deep vein thrombosis

Exclusion Criteria:

* Contraindication to comparator drugs
* Symptomatic Pulmonary embolism
* Conditions with increased bleeding risk
* Unstable patients with reduced life expectancy
* Severe renal impairment
* Impaired liver function
* Strong CYP 3A4 inhibitors
* Platelet aggregation inhibitors (exception: ASA up to 500mg) therapy with anticoagulants or fibrinolytics
* NSAIDs with half-life > 17 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2004-03; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Response to treatment as determined by a Complete Compression Ultra sound (CCUS) | 21 days

SECONDARY OUTCOMES:
Response to treatment as determined by a Complete Compression Ultrasound (CCUS) and perfusion lung scan | Day 21
Response to treatment and residual vein diameter as assessed by Complete Compression Ultrasound (CCUS) | Day 84
Incidence of symptomatic and confirmed recurrence or extension of Deep Vein Thrombosis (DVT) | Day 1-84
Composite endpoint of symptomatic and confirmed recurrence and extension of Deep Vein Thrombosis (DVT) and symptomatic Pulmonary Embolism (PE) (nonfatal DVT and/or nonfatal PE) and deaths during the 3 months treatment period | Day 1-84
Incidence of symptomatic and confirmed recurrence and extension of Deep Vein Thrombosis (DVT) and symptomatic Pulmonary Embolism (PE) within 30 days after stop of treatment with study drug | Day 1-114

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (93):
- Australia (4):
  - Sydney, New South Wales
  - Adelaide, South Australia
  - Melbourne, Victoria
  - Perth, Western Australia
- Austria (2):
  - Graz, Styria
  - Vienna
- Belgium (2):
  - Duffel
  - Leuven
- São Paulo, São Paulo, Brazil
- Canada (9):
  - Vancouver, British Columbia
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - North Bay, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
- Colombia (3):
  - Barranquilla
  - Bogotá
  - Medellín
- Czechia (5):
  - Brno
  - Kladno
  - Ostrava
  - Pilsen
  - Prague
- Germany (9):
  - Heidelberg, Baden-Wurttemberg
  - Karlsbad, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - München, Bavaria
  - Darmstadt, Hesse
  - Bergisch Gladbach, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Dresden, Saxony
  - Berlin
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szentes
- Israel (7):
  - Afula
  - Ashkelon
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Tel Aviv
- Italy (9):
  - Rozzano, Milano
  - Bologna
  - Milan
  - Padua
  - Palermo
  - Perugia
  - Piacenza
  - Reggio Emilia
  - Varese
- Netherlands (7):
  - 's-Hertogenbosch
  - Arnhem
  - Dirksland
  - Enschede
  - Leidschendam
  - Rotterdam
  - The Hague
- New Zealand (2):
  - Auckland
  - Christchurch
- Peru (2):
  - Lima
  - Lima Cercado
- Poland (8):
  - Bialystok
  - Bytom
  - Gdansk
  - Katowice
  - Lublin
  - Olsztyn
  - Poznan
  - Warsaw
- South Africa (4):
  - Bloemfontein, Freestate
  - Pretoria, Gauteng
  - Cape Town, Western Cape
  - Somerset West, Western Cape
- Spain (7):
  - Badalona, Barcelona
  - Olot, Girona
  - San Cristóbal de La Laguna, Tenerife
  - Barcelona
  - Girona
  - Madrid
  - Valencia
- Sweden (4):
  - Gothenburg
  - Halmstad
  - Jönköping
  - Lund
- Switzerland (4):
  - Basel
  - Bern
  - Lucerne
  - Zurich

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu